CLINICAL TRIAL: NCT02535585
Title: Arthroscopic Treatment of Anterior Shoulder Dislocation Using Knotted and Knotless Anchors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Frederico Lafraia Lobo, physician, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1134
Record Dates: First submitted 2015-08-21; First posted 2015-08-28 (Estimated); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Shoulder Dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- knotted anchors (Active Comparator): Arthroscopic repair of the labral lesion with knotted anchors (SutureTak biocomposite 3.0 mm).
  Interventions: Device: knotted anchors (SutureTak biocomposite 3.0 mm)
- knotless anchors (Active Comparator): Arthroscopic repair of the labral lesion with knotless anchors (PushLock biocomposite 2.9 mm knotless)
  Interventions: Device: knotless anchors (PushLock biocomposite 2.9 mm knotless)

INTERVENTIONS:
Device: knotted anchors (SutureTak biocomposite 3.0 mm) — Arthroscopic repair of the labral lesion with knotted anchors (SutureTak biocomposite 3.0 mm).
  Arms: knotted anchors
Device: knotless anchors (PushLock biocomposite 2.9 mm knotless) — Arthroscopic repair of the labral lesion with knotless anchors (PushLock biocomposite 2.9 mm knotless)
  Arms: knotless anchors

SUMMARY:
The shoulder is the joint that most commonly suffers dislocation, and anterior instability is the most frequent form. Arthroscopic repair is the gold standard for the treatment of recurrent shoulder dislocation. The most commonly used technique is the attachment of glenoid labrum-ligament complex (GLLC) with knotted anchors. In 2001, Thal introduced the concept of tissue fixation using knotless anchors and its applicability for GLLC lesions. Some researchers have published studies using knotless anchors and have compared this technique to the use of knotted anchors, demonstrating similar reconstruction of labral height and functional outcomes, while the recurrence rate is still contradictory. To date, there are no prospective randomized controlled clinical trial comparing these two techniques of GLLC repairs.

The researchers aims to compare clinical outcomes and imaging evaluation of patients undergoing GLLC repair arthroscopically with the use of absorbable knotless and knotted anchors.

DETAILED DESCRIPTION:
The shoulder is the joint that most commonly suffers dislocation, and anterior instability is the most frequent form. The overall incidence of first-time dislocations requiring closed reduction is 23.1 per 100,000 people/year, with a higher incidence in males and Caucasians. Individuals with a younger age at first dislocation show a higher rate of recurrence.

Arthroscopic repair is the gold standard for the treatment of recurrent shoulder dislocation, with similar outcomes to open repair. The technique is less aggressive because the tendon of the subscapularis does not need to be addressed, leading to shorter hospital stays, less scarring, earlier return to normal activities, and a greater postoperative range of motion.

In this technique, the glenoid labrum-ligament complex (GLLC) is repaired using bone anchors that can be metallic, absorbable, or flexible. Biomechanical studies have shown that these three types of anchors are similar in terms of cyclic loading resistance and bone fixation. Absorbable anchors are most frequently used because metallic anchors can cause postoperative imaging interference in MRI study, can migrate and became loose or break, which can damage the articular cartilage. Flexible anchors when submitted to cyclic stress can produce cystic cavities in bone tissue attachment 21, and probably can lead to a failure of glenoid labrum-ligament complex suture.

The most commonly used technique is the attachment of GLLC with knotted anchors. Studies have shown to perform an arthroscopic knot is challenging and can be technically difficult. The knot volume can produce friction during the shoulder movement, leading joint discomfort and cartilage damage. The quality of the soft tissue healing depend on the knot quality too. The dislocation recurrence rate with this technique ranges from 4% to 19%.

In 2001, Thal introduced the concept of tissue fixation using knotless anchors and its applicability for GLLC lesions. Although this new technique had solved the difficulty of tying knots, the results regarding the GLLC suture shown more gap formation between this complex and the glenoid bone, delayed anchor loosening and postoperative arthropathy. The recurrence rate is high associated with perianchor radiolucency.The recurrence rate with this technique is as high as 23.8%.

Some researchers have published studies using knotless anchors and have compared this technique to the use of knotted anchors, demonstrating similar reconstruction of labral height and functional outcomes, while the recurrence rate is still contradictory. To date, there are no prospective randomized controlled clinical trial comparing these two techniques of GLLC repairs.

Our researchers aims to compare clinical outcomes and imaging evaluation of patients undergoing GLLC repair arthroscopically with the use of absorbable knotless and knotted anchors.

ELIGIBILITY:
Inclusion Criteria:

* Skeletal maturity;
* Anterior glenohumeral instability;
* Previous labral lesion without bone defects or with defects that affect no more than 20% of the anteroposterior diameter of the glenoid, as shown by MRI;
* Instability severity index score (ISIS) < 4;

Non-Inclusion Criteria

* Epilepsy;
* Associated rotator cuff tear;
* Proximal humeral fracture;
* Multidirectional or posterior instability by clinical evaluation;
* Generalized ligamentous laxity by clinical evaluation;

Exclusion Criteria:

* Irreparable injury to the anterior capsule or injury to the humeral insertion of the inferior glenohumeral ligament;
* Glenoid bone defect greater than 20% of the anteroposterior diameter measured by arthroscopy;
* Rotator cuff tear found on arthroscopy;
* Abandonment of the rehabilitation program and follow-up before the first evaluation of outcomes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2021-01-16 (Actual)

PRIMARY OUTCOMES:
Rowe scale | 1 year
  To compare, using the Rowe scale, clinical outcomes, at one year after surgery, of patients undergoing labral lesion suture using knotted anchors with those treated with knotless anchors.

SECONDARY OUTCOMES:
dislocation recurrence rate | 1 year
  To evaluate the postoperative dislocation recurrence rate in each group of patients
intraoperative and postoperative complications | 1 year
  To ascertain intraoperative (loosening, protrusion, and breaking of material) and postoperative (infection, stiffness, and osteoarthritis) complications
WOSI | 1 year
  To compare the clinical outcomes of the two patient groups using the Western Ontario Shoulder Instability Index (WOSI).
ASES | 1 year
  To compare the clinical outcomes of the two patient groups using the American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES).
Magnetic resonance imaging - LGHI | 1 year
  Labrum glenoid height index (LGHI) - ratio of the labral height to the glenoid height
Magnetic resonance imaging - Labral Slope | 1 year
  Labral slope - angle between the line perpendicular to the deepest point of the glenoid to the labral glenoid apex
Magnetic resonance imaging - Labral morphology | 1 year
  Labral morphology (PDW EXP sequence) with the Rondelli classification
Magnetic resonance imaging - Anchor resorption | 1 year
  Anchor resorption (T1 sequence) according to Stein et al.
Magnetic resonance imaging - Bone reaction | 1 year
  Bone reaction (T2 sequence) according to Hoffmann et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Departamento de Ortopedia e Traumatologia do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Cutts S, Prempeh M, Drew S. Anterior shoulder dislocation. Ann R Coll Surg Engl. 2009 Jan;91(1):2-7. doi: 10.1308/003588409X359123. PMID 19126329
- [Background] Leroux T, Wasserstein D, Veillette C, Khoshbin A, Henry P, Chahal J, Austin P, Mahomed N, Ogilvie-Harris D. Epidemiology of primary anterior shoulder dislocation requiring closed reduction in Ontario, Canada. Am J Sports Med. 2014 Feb;42(2):442-50. doi: 10.1177/0363546513510391. Epub 2013 Nov 25. PMID 24275862
- [Background] Owens BD, Dawson L, Burks R, Cameron KL. Incidence of shoulder dislocation in the United States military: demographic considerations from a high-risk population. J Bone Joint Surg Am. 2009 Apr;91(4):791-6. doi: 10.2106/JBJS.H.00514. PMID 19339562
- [Background] Harris JD, Gupta AK, Mall NA, Abrams GD, McCormick FM, Cole BJ, Bach BR Jr, Romeo AA, Verma NN. Long-term outcomes after Bankart shoulder stabilization. Arthroscopy. 2013 May;29(5):920-33. doi: 10.1016/j.arthro.2012.11.010. Epub 2013 Feb 5. PMID 23395467
- [Background] Bollier MJ, Arciero R. Management of glenoid and humeral bone loss. Sports Med Arthrosc Rev. 2010 Sep;18(3):140-8. doi: 10.1097/JSA.0b013e3181e88ef9. PMID 20711045
- [Background] Kim SH, Ha KI, Cho YB, Ryu BD, Oh I. Arthroscopic anterior stabilization of the shoulder: two to six-year follow-up. J Bone Joint Surg Am. 2003 Aug;85(8):1511-8. PMID 12925631
- [Background] Carreira DS, Mazzocca AD, Oryhon J, Brown FM, Hayden JK, Romeo AA. A prospective outcome evaluation of arthroscopic Bankart repairs: minimum 2-year follow-up. Am J Sports Med. 2006 May;34(5):771-7. doi: 10.1177/0363546505283259. PMID 16627629
- [Background] Burkhart SS, De Beer JF. Traumatic glenohumeral bone defects and their relationship to failure of arthroscopic Bankart repairs: significance of the inverted-pear glenoid and the humeral engaging Hill-Sachs lesion. Arthroscopy. 2000 Oct;16(7):677-94. doi: 10.1053/jars.2000.17715. PMID 11027751
- [Background] Fabbriciani C, Milano G, Demontis A, Fadda S, Ziranu F, Mulas PD. Arthroscopic versus open treatment of Bankart lesion of the shoulder: a prospective randomized study. Arthroscopy. 2004 May;20(5):456-62. doi: 10.1016/j.arthro.2004.03.001. PMID 15122134
- [Background] Hayashida K, Yoneda M, Mizuno N, Fukushima S, Nakagawa S. Arthroscopic Bankart repair with knotless suture anchor for traumatic anterior shoulder instability: results of short-term follow-up. Arthroscopy. 2006 Jun;22(6):620-6. doi: 10.1016/j.arthro.2006.03.006. PMID 16762700
- [Background] Ng C, Bialocerkowski A, Hinman R. Effectiveness of arthroscopic versus open surgical stabilisation for the management of traumatic anterior glenohumeral instability. Int J Evid Based Healthc. 2007 Jun;5(2):182-207. doi: 10.1111/j.1479-6988.2007.00064.x. PMID 21631787
- [Background] Kim SH, Ha KI, Kim SH. Bankart repair in traumatic anterior shoulder instability: open versus arthroscopic technique. Arthroscopy. 2002 Sep;18(7):755-63. doi: 10.1053/jars.2002.31701. PMID 12209434
- [Background] Hobby J, Griffin D, Dunbar M, Boileau P. Is arthroscopic surgery for stabilisation of chronic shoulder instability as effective as open surgery? A systematic review and meta-analysis of 62 studies including 3044 arthroscopic operations. J Bone Joint Surg Br. 2007 Sep;89(9):1188-96. doi: 10.1302/0301-620X.89B9.18467. PMID 17905956
- [Background] Cooke SJ, Starks I, Kathuria V. The results of arthroscopic anterior stabilisation of the shoulder using the bioknotless anchor system. Sports Med Arthrosc Rehabil Ther Technol. 2009 Jan 19;1(1):2. doi: 10.1186/1758-2555-1-2. PMID 19284697
- [Background] Barber FA, Herbert MA. Cyclic loading biomechanical analysis of the pullout strengths of rotator cuff and glenoid anchors: 2013 update. Arthroscopy. 2013 May;29(5):832-44. doi: 10.1016/j.arthro.2013.01.028. Epub 2013 Apr 2. PMID 23561482
- [Background] Mazzocca AD, Chowaniec D, Cote MP, Fierra J, Apostolakos J, Nowak M, Arciero RA, Beitzel K. Biomechanical evaluation of classic solid and novel all-soft suture anchors for glenoid labral repair. Arthroscopy. 2012 May;28(5):642-8. doi: 10.1016/j.arthro.2011.10.024. Epub 2012 Feb 1. PMID 22301360
- [Background] Gaenslen ES, Satterlee CC, Hinson GW. Magnetic resonance imaging for evaluation of failed repairs of the rotator cuff. Relationship to operative findings. J Bone Joint Surg Am. 1996 Sep;78(9):1391-6. doi: 10.2106/00004623-199609000-00015. PMID 8816656
- [Background] Silver MD, Daigneault JP. Symptomatic interarticular migration of glenoid suture anchors. Arthroscopy. 2000 Jan-Feb;16(1):102-5. doi: 10.1016/s0749-8063(00)90136-1. PMID 10627354
- [Background] Rhee YG, Lee DH, Chun IH, Bae SC. Glenohumeral arthropathy after arthroscopic anterior shoulder stabilization. Arthroscopy. 2004 Apr;20(4):402-6. doi: 10.1016/j.arthro.2004.01.027. PMID 15067280
- [Background] Kaar TK, Schenck RC Jr, Wirth MA, Rockwood CA Jr. Complications of metallic suture anchors in shoulder surgery: A report of 8 cases. Arthroscopy. 2001 Jan;17(1):31-7. doi: 10.1053/jars.2001.18246. PMID 11154364
- [Background] Pfeiffer FM, Smith MJ, Cook JL, Kuroki K. The histologic and biomechanical response of two commercially available small glenoid anchors for use in labral repairs. J Shoulder Elbow Surg. 2014 Aug;23(8):1156-61. doi: 10.1016/j.jse.2013.12.036. Epub 2014 Apr 13. PMID 24725901
- [Background] Rhee YG, Ha JH, Cho NS. Anterior shoulder stabilization in collision athletes: arthroscopic versus open Bankart repair. Am J Sports Med. 2006 Jun;34(6):979-85. doi: 10.1177/0363546505283267. Epub 2006 Jan 25. PMID 16436537
- [Background] Mazzocca AD, Brown FM Jr, Carreira DS, Hayden J, Romeo AA. Arthroscopic anterior shoulder stabilization of collision and contact athletes. Am J Sports Med. 2005 Jan;33(1):52-60. doi: 10.1177/0363546504268037. PMID 15610999
- [Background] Ide J, Maeda S, Takagi K. Arthroscopic Bankart repair using suture anchors in athletes: patient selection and postoperative sports activity. Am J Sports Med. 2004 Dec;32(8):1899-905. doi: 10.1177/0363546504265264. PMID 15572319
- [Background] Cho NS, Hwang JC, Rhee YG. Arthroscopic stabilization in anterior shoulder instability: collision athletes versus noncollision athletes. Arthroscopy. 2006 Sep;22(9):947-53. doi: 10.1016/j.arthro.2006.05.015. PMID 16952723
- [Background] Thal R. Knotless suture anchor: arthroscopic bankart repair without tying knots. Clin Orthop Relat Res. 2001 Sep;(390):42-51. PMID 11550875
- [Background] Riboh JC, Heckman DS, Glisson RR, Moorman CT 3rd. Shortcuts in arthroscopic knot tying: do they affect knot and loop security? Am J Sports Med. 2012 Jul;40(7):1572-7. doi: 10.1177/0363546512446676. Epub 2012 May 10. PMID 22582226
- [Background] Loutzenheiser TD, Harryman DT 2nd, Yung SW, France MP, Sidles JA. Optimizing arthroscopic knots. Arthroscopy. 1995 Apr;11(2):199-206. doi: 10.1016/0749-8063(95)90067-5. PMID 7794433
- [Background] Thal R, Nofziger M, Bridges M, Kim JJ. Arthroscopic Bankart repair using Knotless or BioKnotless suture anchors: 2- to 7-year results. Arthroscopy. 2007 Apr;23(4):367-75. doi: 10.1016/j.arthro.2006.11.024. PMID 17418328
- [Background] Sugaya H, Moriishi J, Kanisawa I, Tsuchiya A. Arthroscopic osseous Bankart repair for chronic recurrent traumatic anterior glenohumeral instability. J Bone Joint Surg Am. 2005 Aug;87(8):1752-60. doi: 10.2106/JBJS.D.02204. PMID 16085615
- [Background] Voos JE, Livermore RW, Feeley BT, Altchek DW, Williams RJ, Warren RF, Cordasco FA, Allen AA; HSS Sports Medicine Service. Prospective evaluation of arthroscopic bankart repairs for anterior instability. Am J Sports Med. 2010 Feb;38(2):302-7. doi: 10.1177/0363546509348049. Epub 2009 Dec 22. PMID 20028847
- [Background] Thal R. A knotless suture anchor. Design, function, and biomechanical testing. Am J Sports Med. 2001 Sep-Oct;29(5):646-9. doi: 10.1177/03635465010290051901. PMID 11573925
- [Background] Thal R. A Knotless Suture Anchor: Technique for use in arthroscopic Bankart repair. Arthroscopy. 2001 Feb;17(2):213-8. doi: 10.1053/jars.2001.20666. PMID 11172255
- [Background] Zumstein M, Jacob HA, Schneeberger AG. In vitro comparison of standard and Knotless metal suture anchors. Arthroscopy. 2004 May;20(5):517-20. doi: 10.1016/j.arthro.2004.03.007. PMID 15122142
- [Background] Antonogiannakis E, Yiannakopoulos CK, Karliaftis K, Karabalis C. Late disengagement of a knotless anchor. Arthroscopy. 2002 Oct;18(8):E40. doi: 10.1053/jars.2002.30008. PMID 12368800
- [Background] Park JY, Lhee SH, Park HK, Jeon SH, Oh JH. Perianchor radiolucency after knotless anchor repair for shoulder instability: correlation with clinical results of 69 cases. Am J Sports Med. 2009 Feb;37(2):360-70. doi: 10.1177/0363546508324312. Epub 2008 Oct 20. PMID 18936278
- [Background] Cho NS, Lubis AM, Ha JH, Rhee YG. Clinical results of arthroscopic bankart repair with knot-tying and knotless suture anchors. Arthroscopy. 2006 Dec;22(12):1276-82. doi: 10.1016/j.arthro.2006.07.005. PMID 17157725
- [Background] Garofalo R, Mocci A, Moretti B, Callari E, Di Giacomo G, Theumann N, Cikes A, Mouhsine E. Arthroscopic treatment of anterior shoulder instability using knotless suture anchors. Arthroscopy. 2005 Nov;21(11):1283-9. doi: 10.1016/j.arthro.2005.08.033. PMID 16325077
- [Background] Kocaoglu B, Guven O, Nalbantoglu U, Aydin N, Haklar U. No difference between knotless sutures and suture anchors in arthroscopic repair of Bankart lesions in collision athletes. Knee Surg Sports Traumatol Arthrosc. 2009 Jul;17(7):844-9. doi: 10.1007/s00167-009-0811-3. Epub 2009 Apr 29. PMID 19404611
- [Background] Ng DZ, Kumar VP. Arthroscopic Bankart repair using knot-tying versus knotless suture anchors: is there a difference? Arthroscopy. 2014 Apr;30(4):422-7. doi: 10.1016/j.arthro.2014.01.005. PMID 24680302
- [Background] Slabaugh MA, Friel NA, Wang VM, Cole BJ. Restoring the labral height for treatment of Bankart lesions: a comparison of suture anchor constructs. Arthroscopy. 2010 May;26(5):587-91. doi: 10.1016/j.arthro.2009.09.010. Epub 2010 Mar 4. PMID 20434654
- [Background] Rowe CR, Patel D, Southmayd WW. The Bankart procedure: a long-term end-result study. J Bone Joint Surg Am. 1978 Jan;60(1):1-16. PMID 624747
- [Background] Piasecki DP, Verma NN, Romeo AA, Levine WN, Bach BR Jr, Provencher MT. Glenoid bone deficiency in recurrent anterior shoulder instability: diagnosis and management. J Am Acad Orthop Surg. 2009 Aug;17(8):482-93. doi: 10.5435/00124635-200908000-00002. PMID 19652030
- [Background] Cho SH, Cho NS, Rhee YG. Preoperative analysis of the Hill-Sachs lesion in anterior shoulder instability: how to predict engagement of the lesion. Am J Sports Med. 2011 Nov;39(11):2389-95. doi: 10.1177/0363546511398644. Epub 2011 Mar 11. PMID 21398576
- [Background] Saito H, Itoi E, Minagawa H, Yamamoto N, Tuoheti Y, Seki N. Location of the Hill-Sachs lesion in shoulders with recurrent anterior dislocation. Arch Orthop Trauma Surg. 2009 Oct;129(10):1327-34. doi: 10.1007/s00402-009-0854-4. Epub 2009 Mar 20. PMID 19301017
- [Background] Burkhart SS, Debeer JF, Tehrany AM, Parten PM. Quantifying glenoid bone loss arthroscopically in shoulder instability. Arthroscopy. 2002 May-Jun;18(5):488-91. doi: 10.1053/jars.2002.32212. PMID 11987058
- [Background] Lo IK, Parten PM, Burkhart SS. The inverted pear glenoid: an indicator of significant glenoid bone loss. Arthroscopy. 2004 Feb;20(2):169-74. doi: 10.1016/j.arthro.2003.11.036. PMID 14760350
- [Background] Wolf EM. Anterior portals in shoulder arthroscopy. Arthroscopy. 1989;5(3):201-8. doi: 10.1016/0749-8063(89)90172-2. PMID 2775394
- [Background] Dahl KA, Patton DJ, Dai Q, Wongworawat MD. Biomechanical characteristics of 9 arthroscopic knots. Arthroscopy. 2010 Jun;26(6):813-8. doi: 10.1016/j.arthro.2009.10.011. PMID 20511040
- [Background] Stein T, Mehling AP, Reck C, Buckup J, Efe T, Hoffmann R, Jager A, Welsch F. MRI assessment of the structural labrum integrity after Bankart repair using knotless bio-anchors. Knee Surg Sports Traumatol Arthrosc. 2011 Oct;19(10):1771-9. doi: 10.1007/s00167-011-1407-2. Epub 2011 Feb 11. PMID 21311867
- [Background] Hoffmann R, Weller A, Helling HJ, Krettek C, Rehm KE. [Local foreign body reactions to biodegradable implants. A classification]. Unfallchirurg. 1997 Aug;100(8):658-66. doi: 10.1007/s001130050172. German. PMID 9381215
- [Background] Balg F, Boileau P. The instability severity index score. A simple pre-operative score to select patients for arthroscopic or open shoulder stabilisation. J Bone Joint Surg Br. 2007 Nov;89(11):1470-7. doi: 10.1302/0301-620X.89B11.18962. PMID 17998184
- [Background] Kirkley A, Griffin S, McLintock H, Ng L. The development and evaluation of a disease-specific quality of life measurement tool for shoulder instability. The Western Ontario Shoulder Instability Index (WOSI). Am J Sports Med. 1998 Nov-Dec;26(6):764-72. doi: 10.1177/03635465980260060501. PMID 9850776
- [Background] Michener LA, McClure PW, Sennett BJ. American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form, patient self-report section: reliability, validity, and responsiveness. J Shoulder Elbow Surg. 2002 Nov-Dec;11(6):587-94. doi: 10.1067/mse.2002.127096. PMID 12469084